CLINICAL TRIAL: NCT00294463
Title: Effects of Tibolone Treatment on the Endometrium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Organon (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 217.640/2002/220
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Postmenopause; Osteoporosis
Keywords: postmenopause; endometrium; Gene Expression Profiling; Histology, Comparative; Hormone Replacement Therapy; Hormones
MeSH Terms: conditions — Osteoporosis | interventions — tibolone; Estradiol

INTERVENTIONS:
Drug: Tibolone
Drug: Estradiol
Drug: Estradiol + Medroxy Progesterone Acetate

SUMMARY:
Tibolone, a tissue-selective compound with a combination of estrogenic, progestogenic and androgenic properties, is used as an alternative for estrogen or estrogen plus progesterone hormone therapy for the treatment of symptoms associated with menopause and osteoporosis. The current study compares endometrial histology, biochemistry (hormone levels) and gene-expression profiles after short-term (21-days) treatment with tibolone, to the findings after treatment with estradiol-only (E2) and E2+Medroxyprogesterone Acetate (MPA) in healthy postmenopausal women undergoing hysterectomy for endometrial prolaps.

Since short-term tibolone use results in increased spotting and bleeding but long-term treatment with tibolone has been shown to lead to an atrophic endometrium our hypothesis is that tibolone first displays a more estrogenic mode of action, which over time, is counterbalanced by tibolone's progestagenic properties

DETAILED DESCRIPTION:
Effects of estrogen deficiency in women are climacteric symptoms and bone loss, which can efficiently be treated by substituting with estrogens (1). Unopposed estrogen treatment, however, increases the risk for endometrial hyperplasia and subsequent carcinoma. For example in the HOPE study (Women's Health, Osteoporosis, Progestin, Estrogen study (2, 3)), after two years of treatment with conjugated equine estrogens (0.625mg/day CEE) the rate of hyperplasia went up to 27,7%. When the treatment was combined with MPA (2.5 mg) the incidence of hyperplasia completely disappeared. Thus, the addition of progestagens is necessary for endometrial safety. Progestagen addition (in continuous combined estrogen plus progestin therapy), however, also causes negative side effects like withdrawal bleeding and an increased breast cancer incidence that was recently documented in the Women's Health Initiative (4) and Million Women Study (5).

Tibolone is a tissue-specific compound used for treatment of climacteric complaints and prevention of osteoporosis and does not stimulate the endometrium like estrogens (6). It is converted by steroid metabolizing enzymes in the liver and intestine into three active metabolites: two hydroxy-metabolites: 3a-hydroxy-tibolone and 3b-hydroxy-tibolone (exerting estrogenic effects and in vivo present in significant amounts) and the delta-4-isomer (exerting progestagenic and androgenic effects, and in vivo present in circulation for a relatively short period of time (7)). The estrogenic metabolites are responsible for the effects on hot flushes, vagina and bone.

Tibolone's effects on the endometrium have been studied by a number of investigators (8-14) using transvaginal ultrasound (TVUS) and histology in biopsies after long-term treatment. With ultrasound it was observed that after 6 years of treatment endometrial thickness was slightly increased (p < 0.05, (8)) in tibolone-users compared to controls. Dőren et al. (9) confirmed that tibolone treatment results in a slight increase in endometrial thickness, which was not different from estrogen + norethisterone acetate treatment (E2+NETA). Histology data after tibolone use for more than 3 months, show no change in 90% of the subjects and only in a few cases an endometrial profile was shown which was comparable to the early follicular phase of a normal cycle (15). Even after two years of tibolone use hyperplasia rarely occurs (10).

In a double-blind, randomized controlled trial, Hammar (16) showed that the bleeding and/or spotting episodes in tibolone users in the first months of use were significantly lower than in E2+NETA users, and the authors hypothesized that this was due to a higher progestagenic activity of tibolone on the endometrium compared to the combined treatment. Our in vitro studies show indeed that tibolone can exert a progestagenic effect and that the balance between the progestagenic properties and the estrogenic properties of tibolone takes effect through a different set of genes acting in the same genetic network (17, 18).

In order to investigate whether our cell line data on tibolone action could be confirmed in vivo, and because relatively short-term effects of tibolone and other hormonal treatments in patients have never been described, postmenopausal women were treated for 21 days with tibolone, estrogen-only, or estrogen together with progestagen (estrogen+progestagen). From these women sera were obtained and endometria were removed in order to assess the histological and immunohistochemical, biochemical (hormone levels) and molecular (gene expression) effects of relatively short-term tibolone use (21-days). The overall results may help us to obtain insight in the mechanism of action of tibolone on the human endometrium compared to reference preparations.

Subjects:

This study was designed as a controlled clinical trial. Patients who visited our clinics (Amphia Hospital Breda, Albert Schweitser Hospital Dordrecht, Erasmus University Medical Center Rotterdam, The Netherlands) to undergo vaginal hysterectomy for treatment of prolapse, were eligible to participate in this study. A description of the inclusion and exclusion criteria of the current experiments were documented earlier (19).

The trial was performed in the period before the scheduled surgery. After informed consent, the patients were sequentially assigned to one of the following treatment groups: Control-group (no hormonal treatment); Tibolone-group (2.5 mg tibolone (Livial, N.V. Organon, Oss, The Netherlands) administered orally every day, starting 21 days prior to surgery); E2 group (2 mg of estradiol administered orally every day, starting 21 days prior to surgery); E2+MPA-group (2 mg estradiol + 5 mg MPA administered orally every day, starting 21 days prior to surgery). The investigators were kept blinded to the patient treatments during the analysis. The study protocol was approved by the local ethics committees of the participating hospitals.

1. van der Mooren MJ, Kenemans P. Postmenopausal Hormone Therapy: Impact on Menopause-Related Symptoms, Chronic Disease and Quality of Life. Drugs 2004;64:821-836.
2. Pickar JH, Yeh I, Wheeler JE, Cunnane MF, Speroff L. Endometrial effects of lower doses of conjugated equine estrogens and medroxyprogesterone acetate. Journal Article. Multicenter Study. Randomized Controlled Trial] Fertil Steril 2001;76:25-31.
3. Pickar JH, Yeh IT, Wheeler JE, Cunnane MF, Speroff L. Endometrial effects of lower doses of conjugated equine estrogens and medroxyprogesterone acetate: two-year substudy results. Fertil Steril 2003;80:1234-40.
4. Anderson GL, Judd HL, Kaunitz AM, Barad DH, Beresford SA, Pettinger M, Liu J, McNeeley SG, Lopez AM; for the Women's Health Initiative Investigators. Effects of estrogen plus progestin on gynecologic cancers and associated diagnostic procedures: the Women's Health Initiative randomized trial. JAMA 2003;290:1739-1748.
5. Beral V, Million Women Study Collaborators. Breast cancer and hormone- replacement therapy in the Million Women Study. Lancet 2003;362:419-27.
6. Kloosterboer HJ. Tibolone: a steroid with a tissue-specific mode of action. J Steroid Biochem Mol Biol 2001;76:231-8.
7. Timmer CJ, Verheul HA, Doorstam DP. Pharmacokinetics of tibolone in early and late postmenopausal women. Br J Clin Pharmacol 2002;54:101-6.
8. Morris EP, Wilson PO, Robinson J, Rymer JM. Long term effects of tibolone on the genital tract in postmenopausal women. Br J Obstet Gynaecol 1999;106:954-9.
9. Dőren M, Rubig A, Coelingh Bennink HJ, Holzgreve W. Impact on uterine bleeding and endometrial thickness: tibolone compared with continuous combined estradiol and norethisterone acetate replacement therapy. Menopause 1999;6:299-306.
10. Volker W, Coelingh Bennink HJ, Helmond FA. Effects of tibolone on the endometrium. Climacteric 2001;4:203-8.
11. Wender MC, Edelweiss MI, Campos LS, de Castro JA, Spritzer PM. Endometrial assessment in women using tibolone or placebo: 1-year randomized trial and 2-year observational study. Menopause 2004;11:423-9.
12. Botsis D, Kassanos D, Kalogirou D, Antoniou G, Vitoratos N, Karakitsos P. Vaginal ultrasound of the endometrium in postmenopausal women with symptoms of urogenital atrophy on low-dose estrogen or tibolone treatment: a comparison. Maturitas 1997;26:57-62.
13. Egarter C, Huber J, Leikermoser R, Haidbauer R, Pusch H, Fischl F, Putz M. Tibolone versus conjugated estrogens and sequential progestogen in the treatment of climacteric complaints. Maturitas 1996;23:55-62.
14. Rymer J, Fogelman I, Chapman MG. The incidence of vaginal bleeding with tibolone treatment. Br J Obstet Gynaecol 1994;101:53-6.
15. Genazzani AR, Benedek-Jaszmann LJ, Hart DM, Andolsek L, Kicovic PM, Tax L. Org OD 14 and the endometrium. Maturitas 1991;13:243-51.
16. Hammar M, Christau S, Nathorst-Boos J, Rud T, Garre K. A double-blind, randomised trial comparing the effects of tibolone and continuous combined hormone replacement therapy in postmenopausal women with menopausal symptoms.Br J Obstet Gynaecol 1998;105:904-11.
17. Blok LJ, De Ruiter PE, Kuhne EC, Hanekamp EE, Grootegoed JA, Smid-Koopman E, Gielen SC, De Gooyer ME, Kloosterboer HJ, Burger CW. Progestogenic effects of tibolone on human endometrial cancer cells. J Clin Endocrinol Metab 2003;88:2327-34.
18. Hanifi-Moghaddam P, Gielen SCJP, Kloosterboer HJ, De Gooyer ME, Sijvers AM, van Gool AJ, Smid M, Morehouse M, Van Wijk FH, Burger CW, Blok LJ. Molecular portrait of the estrogenic and progestagenic actions of tibolone: Behavior of biological networks in response to tibolone. J Clin Endocrinol Metab 2005;90:973-83.
19. Klaassens AHA, Van Wijk FH, Hanifi-Moghaddam P, Sijmons B, Ewing PC, Ten Kate-Booij MJ, Kooi GS, Kloosterboer HJ, Blok LJ, Burger CW. Histological and immunohistochemical evaluation of postmenopausal endometrium after 3 weeks of treatment with tibolone, estrogen-only, or estrogen plus progestagen. Accepted in Fertility and Sterility, 2006

ELIGIBILITY:
Inclusion Criteria:

Healthy postmenopausal women with a uterus. "Postmenopausal'' was defined as amenorrhoeic for at least one year prior to screening, or amenorrhoeic for at least six months prior to screening with a serum E2 concentration of < 20 pg/ml and a serum FSH concentration of > 40 IU/L at screening. If the patient used any kind of steroid hormone therapy prior to the study, a washout period of 6 months (for intra-uterine progesterone and oral estrogen+progestagen combination therapy) or 12 months (for progesterone implants or injections and injected estrogen+progestagen combination therapy) was applied.

Exclusion Criteria:

1. Histological diagnosis by a local pathologist of an endometrial biopsy (with the Pipelle suction curette) taken before treatment, as proliferative, secretory or menstrual type endometrium, endometrial metaplasia, endometrial or endocervical polyp(s), endometrial hyperplasia, cancer or any other histological abnormality (leiomyoma(ta), stromal nodules or mesenchymal or (endo)cervical neoplasia(s)).
2. Double-layer endometrium thickness > 4 mm as assessed by transvaginal ultrasound, immediately before endometrial biopsy.
3. History or presence of any malignancy, except successfully treated non-melanoma skin cancers.
4. Any unexpected vaginal bleeding following the menopause.
5. Liver disease, except cholecystectomy.
6. Abnormal cervical Pap smear test result, or abnormal mammography result obtained within one year prior to the start of the trial
7. Deep vein thrombosis, thrombophlebitis, thromboembolic disease, or suspicions of having hereditary predisposition for developing venous thromboembolic disease.
8. Use of one or more of the following drugs within the last two months: hepatic microsomal enzyme-inducing anticonvulsant drugs known to affect or interfere with the pharmacokinetics of steroids (e.g. hydantoins, barbiturates such as Phenobarbital (alone or in combinations, such as Bellergal) rifampicin, griseofulvin, primidone or carbamazepine).

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2003-02; Study Completion 2005-03

PRIMARY OUTCOMES:
Histologic evaluation of the endometrium at the end of treatment
Biochemical evaluation (hormone measurements) of uterine tissue at the end of treatment
Biochemical evaluation of sera, obtained just prior to treatment and at surgery
Molecular assessment of gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Curt W Burger, MD, PhD, Principal Investigator — Erasmus MC, P.O. Box 2040, 3000 CA Rotterdam, The Netherlands; Leen J Blok, PhD, Principal Investigator — Erasmus MC, P.O. Box 2040, 3000 CA Rotterdam, The Netherlands
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Derived] Hanifi-Moghaddam P, Boers-Sijmons B, Klaassens AH, van Wijk FH, Van Ijcken WF, Van der Spek P, Verheul HA, Kloosterboer HJ, Burger CW, Blok LJ. Difference in signalling between various hormone therapies in endometrium, myometrium and upper part of the vagina. Hum Reprod. 2008 Feb;23(2):298-305. doi: 10.1093/humrep/dem366. Epub 2007 Dec 11. PMID 18077316